CLINICAL TRIAL: NCT05627336
Title: Causes and Frequency of Tokophobia, Its Effect on Cesarean Delivery Rates: Our Clinical Experience
Brief Title: Tokophobia ; Our Clinical Experience
Status: Active, not recruiting | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Pinar KADIROGULLARI Assoc.Prof, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ATADEK/ 11.2022
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Tocophobia; Pregnancy Complications
Keywords: vaginal birth; cesarean delivery; fear of childbirth
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: pregnant women in the 3rd trimester — Pregnant women who are in their third trimester and will give birth in the clinic will form the study group. These pregnant women will be measured by applying a set of questionnaires to measure their fear of childbirth.

SUMMARY:
Fear of childbirth, or what has historically been called tokophobia, is often described as a severe fear of birth and pathological fear of childbirth. The reasons for fear of childbirth are stated as biological reasons, psychological reasons and lack of social support. However, it is still not possible to clearly explain the reasons for the fear of childbirth in pregnant women and the risk factors affecting them. The reasons for the fear of childbirth and the affecting factors have not been fully explained.

DETAILED DESCRIPTION:
The aim of this study is to examine the relationship between fear of childbirth and anxiety sensitivity in pregnant women, and whether the mode of delivery changes depending on this fear and these data. The aim of the authors is to reveal the frequency and causes of tokophobia in pregnant women followed in their clinics and to show the birth patterns of these patients.

ELIGIBILITY:
Inclusion Criteria:

* 3rd trimester pregnant women who are followed up in our clinic and will give birth in our clinic.
* Pregnant women between the ages of 18 and 40

Exclusion Criteria:

* Those in the risky pregnancy category (preeclampsia, gdm, iugr… etc.)
* Known to have fetal anomaly during follow-ups
* Those with chronic disease
* Those with sexually transmitted diseases
* Those with a history of cesarean section

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female pregnant women
Study Population: 3rd trimester pregnant women who are followed up in our clinic and will give birth in our clinic. Pregnant women between the ages of 18 and 40
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
diagnosis of tokophobia | 2 months
  patients will be administered W-DEQ: Wijma Delivery Expectancy/Experience Questionnaire part A. As a result, those who score above 85 will be diagnosed with tokophobia.
  this test; Each question has a point equivalent, and the diagnosis will be reached by adding all the points at the end.
type of birth | 2 months
  The birth types of patients diagnosed with tokophobia will be examined. It will be tried to show statistically whether tokophobia increases cesarean section rates or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem University Atakent Hospital, Department of Obstetrics and Gynecology,, Istanbul, Turkey (Türkiye)